CLINICAL TRIAL: NCT06709625
Title: Comparison of the Effects of Erector Spinae Plane Block and Transversus Thoracis Muscle Plane Block on Postoperative Recovery in Patients Undergoing Coronary Artery Surgery
Brief Title: Comparison of Erector Spinae Plane Block and Transversus Thoracic Muscle Plane Block in Coronary Artery Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NigarAltindag1
Record Dates: First submitted 2024-02-12; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Nerve Block; Coronary Artery Bypass; Anesthesia and Analgesia
Keywords: Erector spina plane block; Transversus thoracic plane block; Cardiothoracic surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Group 1 patients will undergo bilateral erector spinae plane block. Heart rate (beats/min) and systolic arterial pressure (mmHg) will be measured before and after induction, after skin incision, after sternotomy, 30 minutes after weaning from CPB, and after sternum closure. VAS and BPS will be used to evaluate pain at 0, 4, 8, 12, 24 hours postoperatively.
  Group 2 patients will undergo transversus thoracic plane block and the same parameters as group 1 will be saved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of patients who underwent erector spinae plane block (Active Comparator): 20 ml %0.25 bupivacaine solution will be given under the erector spinae muscle under USG guidance in the prone position and intraoperative and postoperative data will be recorded.
  Interventions: Procedure: Erector spina plane block (ESP)
- Group of patients who undervent transversus thoracic plane block (Active Comparator): 20ml %0.25 bupivacaine solution will be given between the transversus thoracis muscle and the internal intercostal muscle under USG guidance in the supin position and intraoperative and postoperative data will be recorded.
  Interventions: Procedure: Transversus thoracis plane block

INTERVENTIONS:
Procedure: Transversus thoracis plane block — Transversus thoracis plane block will be applied to provide postoperative analgesia.
  Arms: Group of patients who undervent transversus thoracic plane block
Procedure: Erector spina plane block (ESP) — Erector spina plane block will be applied to provide postoperative analgesia.
  Arms: Group of patients who underwent erector spinae plane block

SUMMARY:
The main objective of this study is to evaluate postoperative pain intensity comparatively between erector spinae plane block and transversus thoracic muscle plane block in patients undergoing open coronary artery surgery. The primary question it aims to address is which of these two regional techniques causes less postoperative pain.

DETAILED DESCRIPTION:
Primary aim in this study is to evaluate the postoperative pain severity of erector spina plane block in comparison with transversus thorasis muscle plane block in patients undergoing open coronary artery surgery. Secondary aim is to retrospectively evaluate the analgesic requirements, complications, extubation times, mortality and morbidity of these patients.

The study will be designed as a prospective randomized controlled trial. After ethics committee approval is obtained, the regional anesthesia method to be applied to 60 patients who are planned to undergo coronary artery surgery in the TR Ministry of Health Ankara City Hospital Cardiovascular Surgery Operating Room and who do not have exclusion criteria will be determined according to the closed envelope method, erector spina plan and transversus thorasis muscle plan (two groups) and will be reported to the anesthesiologist.

Patients who will undergo bilateral erector spinae plane block will be taken to the operating room non-premedicated. In the operating room, after ASA monitoring, intra-arterial, BIS, NIRS monitoring, anesthesia induction with propofol 1-3 mg/kg, fentanyl 2 µg/kg and rocuronium 0.6 mg/kg, endotracheal intubation will be performed, central vein catheterization, urinary catheter and nasopharyngeal temperature probe will be placed. . After the patient is placed in the prone position by the same experienced researcher, appropriate sterilization conditions for the skin and equipment are provided, the USG probe will be fixed on the transverse process in the area where the block is desired, and a 22 gauge 80 mm block needle will be placed parallel to the longitudinal axis. The bone structure will be reached by viewing the needle with an in plane technique at an angle of approximately 45 degrees and advancing it to the posterior of the transverse process. When the needle tip is in the appropriate position under the erector spinae muscle, intermittent aspiration will be performed to confirm that there is no vascular puncture. Following negative aspiration, saline is administered and local anesthetic injection is applied after the erector spinae muscle is seen to be separated from the transverse process. For TTP, the same experienced practitioner places the USG probe, which should be placed approximately 2-3 cm lateral to the sternal border, under the same sterile conditions. The T4-T5 intercostal space will then be identified under ultrasound guidance in a parasagittal view, and the nerve block needle is inserted in-plane into the catheter. The needle is then directed into the transversus thoracic muscle plane between this muscle and the internal intercostal muscle. Here, the local anesthetic solution will be given, taking care to aspirate before each injection to avoid intravascular and intrapleural administration.

Anesthesia will be maintained with propofol/oxygen/air mixture and remifentanil 1 mcg/kg/hour. If systolic arterial blood pressure or heart rate increases more than 20% above baseline in response to surgical stimuli, additional fentanyl 2 µg/kg increments will be administered.

IV tramadol PCA bolus 10mg will be prepared for each patient with a lock-in time of 20 minutes and its use will be explained to the patients in the preoperative period. The total dose of madol used will be monitored.

At the end of the surgery, patients will be taken to intensive care and monitored on a mechanical ventilator. According to standard ICU policy, extubation will be performed at the earliest clinically appropriate time. Patients will be monitored in intensive care for 24 hours after extubation. In the ICU, VAS and BPS will be used to evaluate pain. When VAS is greater than 4 and BPS is greater than 3, additional analgesia will be given.

Induction and maintenance anesthetic drugs and dosages, analgesic drugs and dosages (15mg/kg every 8 hours after routine paracetamol, analgesic need with PCA device, total doses, before and after anesthesia induction, after skin incision, after sternotomy, after 30 hours after leaving CPB Minutes later and after closing the sternum, heart rate (beats/min) and systolic arterial pressure (mmHg) will be measured. 0, 4, 8, 12, 24 hours after postoperative extubation, respiratory rate (respiratory rate/min) and from ICU arrival to endotracheal extubation. Extubation time (minutes) defined as the time from extubation to first rescue analgesia (hours), pain problems: time from extubation to first rescue analgesia (hours), VAS and BPS scores at 0, 4, 8, 12, 24 hours after extubation, postoperative pain at rest and sternal Complications associated with the non-pain block will be recorded.

Sample size calculation was performed using MedCalc 15.8 (MedCalc Software bvba, Ostend, Belgium). It was determined that a minimum 60 patient (30+30) was sufficient for 90% (1-β) power.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 who will undergo elective coronary artery surgery in TR Ankara City Hospital cardiovascular surgery operating room will be included in the study.

Exclusion Criteria:

* Exclusion criteria for patients aged 18-80 who will undergo isolated coronary artery bypass surgery
* Non-coronary artery surgery cases
* Re-operations
* Low EF (<40%)
* psychiatric illness
* Those who have contraindications for block (infection at the block site, etc.)
* Patients who do not or cannot give consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the postoperative pain intensity of erector spinae plane block in comparison with transversus thoracis muscle plane block in patients undergoing open coronary artery surgery. | postoperatively 0, 4, 8, 12 and 24 hours
  VAS values will be recorded
To evaluate the postoperative pain intensity of erector spinae plane block in comparison with transversus thoracis muscle plane block in patients undergoing open coronary artery surgery. | postoperatively 0, 4, 8, 12 and 24 hours
  BPS values will be recorded
To evaluate the postoperative pain intensity of erector spinae plane block in comparison with transversus thoracis muscle plane block in patients undergoing open coronary artery surgery. | postoperatively 0, 4, 8, 12 and 24 hours
  Rescue analgesic dosages will be recorded
To evaluate the effects of erector spinae plane block on postoperative hemonidamy in patients undergoing open coronary artery surgery, in comparison with transversus thoracis muscle plane block. | postoperatively 0, 4, 8, 12 and 24 hours
  Systolic arterial pressure will be recorded

SECONDARY OUTCOMES:
Determine the incidence of block-related adverse events | Neurological or cardiovascular events occurring within the first 30 minutes after block application will be monitored to evaluate local anesthesia toxicity.
Determine the incidence of block-related adverse events | Chest wall hematoma and pneumothorax are diagnosed by USG after block and before skin incision within the first 24 hours after block applications
To record the incidence of other side effects due to opioid administration | Postoperatively 0, 2, 4, 8, 12, 24 hours
  t will be questioned whether there is itching or not
To record the incidence of other side effects due to opioid administration | Postoperatively 0, 2, 4, 8, 12, 24 hours
  t will be questioned whether there is nausea or not
To record the incidence of other side effects due to opioid administration | Postoperatively 0, 2, 4, 8, 12, 24 hours
  t will be questioned whether there is vomiting or not
Evaluation of intraoperative hemodynamic changes between two blocks | Heart rate (beats/min) will be measured before and 1minute later after anesthesia induction, 1minute later after skin incision, 1minute later after sternotomy, 30 minutes after weaning from CPB, and 1minute later after sternum closure.
Evaluation of intraoperative hemodynamic changes between two blocks | Before and 1minute later after anesthesia induction, 1minute later after skin incision, 1minute later after sternotomy, 30 minutes after weaning from CPB, and 1minute later after sternum closure.
  Systolic arterial pressure (mmHg) will be measured before and after anesthesia induction, after skin incision, after sternotomy, 30 minutes after weaning from CPB, and after sternum closure.

CONTACTS AND LOCATIONS:
Overall Officials: Nevriye Salman, Principal Investigator — ankara bilkent city hospital, anesthesiology and reanimation clinic
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Result] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Result] Zubrzycki M, Liebold A, Skrabal C, Reinelt H, Ziegler M, Perdas E, Zubrzycka M. Assessment and pathophysiology of pain in cardiac surgery. J Pain Res. 2018 Aug 24;11:1599-1611. doi: 10.2147/JPR.S162067. eCollection 2018. PMID 30197534
- [Result] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Result] Barr LF, Boss MJ, Mazzeffi MA, Taylor BS, Salenger R. Postoperative Multimodal Analgesia in Cardiac Surgery. Crit Care Clin. 2020 Oct;36(4):631-651. doi: 10.1016/j.ccc.2020.06.003. Epub 2020 Aug 12. PMID 32892818
- [Result] Cosarcan SK, Sezer OA, Gurkahraman S, Ercelen O. Regional analgesia techniques for effective recovery from coronary artery bypass surgeries: a retrospective study involving the experience of a single center. J Cardiothorac Surg. 2022 Jul 6;17(1):170. doi: 10.1186/s13019-022-01923-6. PMID 35794614
- [Result] Gregory AJ, Grant MC, Manning MW, Cheung AT, Ender J, Sander M, Zarbock A, Stoppe C, Meineri M, Grocott HP, Ghadimi K, Gutsche JT, Patel PA, Denault A, Shaw A, Fletcher N, Levy JH. Enhanced Recovery After Cardiac Surgery (ERAS Cardiac) Recommendations: An Important First Step-But There Is Much Work to Be Done. J Cardiothorac Vasc Anesth. 2020 Jan;34(1):39-47. doi: 10.1053/j.jvca.2019.09.002. Epub 2019 Sep 7. No abstract available. PMID 31570245
- [Result] King M, Stambulic T, Hassan SMA, Norman PA, Derry K, Payne DM, El Diasty M. Median sternotomy pain after cardiac surgery: To block, or not? A systematic review and meta-analysis. J Card Surg. 2022 Nov;37(11):3729-3742. doi: 10.1111/jocs.16882. Epub 2022 Sep 13. PMID 36098374
- [Result] Cogan J. Pain management after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2010 Sep;14(3):201-4. doi: 10.1177/1089253210378401. PMID 20705642
- [Result] Ritter MJ, Christensen JM, Yalamuri SM. Regional Anesthesia for Cardiac Surgery: A Review of Fascial Plane Blocks and Their Uses. Adv Anesth. 2021 Dec;39:215-240. doi: 10.1016/j.aan.2021.08.001. Epub 2021 Oct 1. No abstract available. PMID 34715976
- [Result] Kelava M, Alfirevic A, Bustamante S, Hargrave J, Marciniak D. Regional Anesthesia in Cardiac Surgery: An Overview of Fascial Plane Chest Wall Blocks. Anesth Analg. 2020 Jul;131(1):127-135. doi: 10.1213/ANE.0000000000004682. PMID 32032103
- [Result] Dost B, De Cassai A, Balzani E, Tulgar S, Ahiskalioglu A. Effects of ultrasound-guided regional anesthesia in cardiac surgery: a systematic review and network meta-analysis. BMC Anesthesiol. 2022 Dec 29;22(1):409. doi: 10.1186/s12871-022-01952-7. PMID 36581838